CLINICAL TRIAL: NCT07284316
Title: Effect of a Multidomain Intervention Plus Turmeric on the Prevention of Cognitive Decline in People Over 55 Years of Age With Insulin Resistance: A Randomized Clinical Trial
Brief Title: Effect of a Multidomain Intervention Plus Turmeric on the Prevention of Cognitive Decline in People Over 55 Years of Age With Insulin Resistance.
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Carlos Arturo Hernández Esquivel, Research, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R-2024-785-058; R-2024-785-058 (Registry Identifier: Effect of a multidomain intervention plus turmeric on the prevention of cognitive decline in people over 55 years of ag)
Record Dates: First submitted 2025-02-18; First posted 2025-12-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Decline; Subjective Cognitive Impairment; Insulin Resistance
Keywords: Subjective cognitive decline; Insulin resistance; Elderly; Multidomain intervention
MeSH Terms: conditions — Cognitive Dysfunction; Insulin Resistance | interventions — turmeric extract; Gelatin

STUDY DESIGN:
Intervention Model Description: To compare the efficacy of a multidomain program (MeMo-Health-Cog-4) with 500 mg/day of turmeric plus 5 mg of black pepper for 24 weeks against a multidomain program (MeMo-Health-Cog-4) with a placebo for the improvement of insulin resistance, global cognitive function (subjective and objective), specific cognitive function (executive function/mental flexibility, verbal learning and memory, and verbal fluency), motor function (gait speed, grip strength, balance, and rising from a chair); reduction of biomarkers of inflammation (IL-6, TNF-alpha, IL-10), endothelial dysfunction (ICAM-1, E-selectin, VCAM-1), and oxidative stress (MDA, GSH) in people aged 55-70 years with insulin resistance; as well as the post-intervention effect at 28 weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The researchers will use key-labeled bottles to designate placebo vs turmeric; the participants, doctors, and staff do not know which group each bottle corresponds to. Only two people from the research team know which group each bottle corresponds to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 500mg capsule grenadine every 12 hours. Measurement of insulin resistance, global cognitive function (subjective and objective), specific cognitive function (executive function/mental flexibility, verbal learning and memory, and verbal fluency), motor function (gait speed, grip strength, balance, and rising from a chair); reduction of biomarkers of inflammation (IL-6, TNF-α, IL-10), endothelial dysfunction (ICAM-1, E-selectin, VCAM-1), and oxidative stress (MDA, GSH) in people aged 55-70 years with insulin resistance; as well as the post-intervention effect at 28 weeks.
  Interventions: Other: Control: Placebo. 500mg gelatin in capsules 2 times a day
- Turmeric extract intervention (Experimental): Multidomain program (MeMo-Health-Cog-4) with 500 mg/day of turmeric plus 5 mg of black pepper for 24 weeks against a multidomain program (MeMo-Health-Cog-4) with a placebo for the improvement of insulin resistance, global cognitive function (subjective and objective), specific cognitive function (executive function/mental flexibility, verbal learning and memory, and verbal fluency), motor function (gait speed, grip strength, balance, and rising from a chair); reduction of biomarkers of inflammation (IL-6, TNF-α, IL-10), endothelial dysfunction (ICAM-1, E-selectin, VCAM-1), and oxidative stress (MDA, GSH) in people aged 55-70 years with insulin resistance; as well as the post-intervention effect at 28 weeks.
  Interventions: Dietary Supplement: Turmeric extract

INTERVENTIONS:
Dietary Supplement: Turmeric extract — The intervention group includes aerobic exercise and cognitive exercise (grid mat), nutritional guidance, a healthy aging program, turmeric capsules, and black pepper
  Arms: Turmeric extract intervention
Other: Control: Placebo. 500mg gelatin in capsules 2 times a day — The control group includes an aerobic exercise program and cognitive exercise (grid mat with various patterns of complexity, applied by a health professional), nutritional guidance, and healthy aging program, plus a placebo.
  Arms: Placebo

SUMMARY:
Introduction: The Insulin resistance itself has been recognized as an independent risk factor for dementia development. Insulin plays an important role in the regulation of muscle function and the processes of learning and memory. Insulin resistance is associated with increased inflammation and oxidative stress. These processes are involved in the pathophysiology of neurodegenerative diseases. Thus, reducing IR could have implications for improving metabolism, muscle, and cognitive function.

Methods and analysis. The investigators will conduct a randomized, double-blind, placebo-controlled clinical trial in which a multidomain program, including an aerobic and cognitive exercise program, will be evaluated. The latter is an exercise program conducted on a checkered mat and will be randomized to participants receiving turmeric plus black pepper or placebo. Participants are affiliated with the Mexican Social Security Institute (IMSS) and are between 55 and 74 years old. The program will last for 24 weeks; after 52 weeks, it will be repeated. The outcomes that the investigators will evaluate are: global cognitive function, specific cognitive function, and the investigators will evaluate serum markers of inflammation, oxidative stress, and GSK-3beta levels. The effect of the interventions on each variable will be analyzed by ANOVA, and a multivariate analysis study with multiple linear regression will be conducted.

Ethics and dissemination of the study: the study was approved by the IMSS National Ethics and Research Committee all participants provided written informed consent prior to their participation.

DETAILED DESCRIPTION:
Dementia is characterized by cognitive impairment, which affects independence in activities of daily living (1). Worldwide, approximately 47 million people were living with dementia in 2015, and before the COVID-19 pandemic, the number of cases was expected to triple by 2050 (2). The prevalence of dementia in Latin America and the Caribbean is 10.66%, and dementia is more prevalent in women than men (7.26%).

Observational studies have shown that dementia and cognitive decline can be prevented by reducing vascular risks and improving healthier lifestyles (6). The key is to modify lifestyle habits before the development of disease symptoms. To achieve this, it is important to characterize populations with intact cognitive function or with some concern without symptoms of cognitive decline (6).

Interventions to treat dementia have been nonpharmacological, including nutrition, cognitive stimulation, physical exercise, and multi-domain (combination of more than two components or domains). However, the best results for dementia prevention have been for multi-domain interventions in individuals with intact cognitive function or those with some concerns (10). The domains included in all multi-domain interventions were physical activity, nutrition, and cognitive training. The Mind and Movement for Cognitive Health Program (MeMo Health-Cog) is a program that includes three basic components: a) a moderate physical activity routine through a one-hour/day routine of combined aerobic exercises, b) cognitive training with the checkered mat and c) a motivational educational program that consists of weekly talks on topics of healthy active aging, sports for older adults, basic nutrition recommendations, health topics, and socialization; these talks last between 10 and 15 minutes. Physical and cognitive activities are a one-hour routine each day, and they can be performed three days a week. The duration of the entire program is 24 weeks. It is important to mention that the educational program encourages light physical activities with the 24-hour healthy educational program, which are recommendations of Canadian origin that allow improving behaviors related to movement, that is, moderate and light physical activities, adequate sleep duration, and limitations of sitting (13).

An important and emerging concept is insulin resistance at the brain level, where insulin signaling plays crucial roles in physiology and therefore affects cognitive function. Altered insulin signaling in brain tissue contributes to Alzheimer's disease (AD) through increased beta-amyloid and tau neurofibrillary tangle formation and other brain damage mechanisms. Insulin resistance not only affects systemic metabolism and directly influences the brain by altering insulin-related brain pathways (20).

b. Mechanisms of insulin resistance, inflammation, and oxidative stress The molecular mechanisms of type 2 diabetes (T2DM) are characterized by an alteration in the regulation of carbohydrate, lipid, and protein metabolism, as a consequence of a decrease in insulin secretion and resistance to its effect (21).

Insulin Resistance (IR). Insulin is a major regulator of carbohydrate, lipid, and protein metabolism. It acts through a signaling cascade involving the receptor, substrate, and various signaling molecules (22, 23). Insulin resistance is defined as an inappropriate response to insulin-mediated glucose control. The skeletal muscle is a quantitatively central tissue for insulin-stimulated glucose disposal, and liver and adipose tissue are qualitatively critical sites for glucose-induced insulin signaling. These tissues are central to understanding the mechanisms responsible for insulin resistance.

Inflammation and oxidative stress are associated with the alteration of insulin signaling, which increases IR. In turn, IR increases oxidative stress and therefore inflammation. Forming a systemic loop of insulin resistance, inflammation and oxidative stress is present in obesity, diabetes, vascular dementia, and Alzheimer's disease (AD); since it affects the function of various organs such as the liver (increases gluconeogenesis), muscle (decreases glucose consumption and loss of muscle mass), adipose tissue (increases adipose tissue), brain (increases neurodegeneration and reduces brain resilience) and cardiovascular system (endothelial dysfunction and vascular damage) (26).

Oxidative stress and insulin resistance (IR). Inflammation promotes oxidative stress and insulin resistance and can also increase GSK-3β expression and alter mitochondrial function, which in turn generate reactive oxygen species (ROS) and nitrogen species (RNS), which react with lipids, proteins and nucleic acids, causing their oxidation and generating neurotoxic consequences (33). Lipid peroxidation, one of the main forms of damage associated with oxidative stress, affects brain tissue and is an important marker of neuronal damage. This damage can be measured by the formation of malondialdehyde (MDA) and 4-hydroxynonenal (HNE), and has been established as a clear factor associated with Alzheimer's disease (AD) (35). In addition, other markers of oxidative stress, such as glutathione levels, are correlated with mild cognitive impairment and AD (36). Other methods to assess oxidative stress include the measurement of protein oxidation, which analyzes the formation of quinones. The accumulation of beta-amyloid (Aβ) plaques and phosphorylated Tau protein in people with type 2 diabetes (T2DM) is associated with inflammation, oxidative stress and insulin resistance (37). At the brain level, insulin reduces the activity of the action of GSK3-β (glycogen synthase kinase-3 beta) as part of its intracellular signaling. This enzyme phosphorylates Tau protein and promotes the division of amyloid precursor protein (APP), and increases the expression of the enzyme BACE-1, resulting in an increase in the amount of beta-amyloid and greater expression of NF-κB

Another function of insulin in the brain is to facilitate brain plasticity, which favors memory and learning by promoting the formation of dendritic spines and synapses; insulin contributes to repair and neuro-protection processes (43)

Since ancient times, functional foods and exercise have been combined to reduce aging-related diseases (49). Dietary choices should have neuroprotective effects. Supplements can cause alterations in signaling pathways, such as AKT, which are important for preventing neurodegeneration because AKT inhibits the activity of GSK-3β, the main enzyme that phosphorylates Tau. Several plants and fruits have shown promise in reducing the progression or risk of dementia, and among the research, curcumin stands out (50). Turmeric is a herbaceous plant whose root, known as rhizome, has been traditionally used both as a spice and for medicinal purposes. Curcuminoids isolated from this plant have anti-inflammatory and immunomodulatory properties.

The main effects attributed to turmeric on health include:

1. Antioxidant effect: it increases the activity of enzymes such as catalase, superoxide dismutase (SOD), glutathione peroxidase and heme-oxygenase (53).
2. Chronic anti-inflammatory effects have been demonstrated in animal studies where it has been shown that inflammation is reduced by decreasing TNF-α levels and suppressing NF-κB activation, as well as by decreasing the expression of inflammatory enzymes such as iNOS, COX-2, lipoxygenase and xanthine oxidase (55). This process reduces the expression of inflammatory cytokines such as IL-1β, IL-6, IL-5, IL-4 and IL-2.
3. Likewise, neuroprotective effects have been observed in animal studies, where turmeric has been shown to inhibit the formation of β-amyloid oligomers and β-amyloid aggregation, in addition to reducing tau hyperphosphorylation. A reduction in neuroinflammation and acetylcholinesterase (AChE) activity was also observed, which could improve memory (56, 57, 58, 59).
4. Regulation of GSK-3β: Studies in mice and clinical trials in humans have shown that curcumin can reduce GSK-3β activity, which may have beneficial effects on insulin resistance and lowering insulin levels (60,53), with this being the only randomized clinical trial that applied 500 mg/day of turmeric for 24 weeks, but improvement in cognitive function has not yet been considered.

Study hypothesis:

The multidomain intervention (MeMo-Health-Cog) with turmeric dietary supplement is more effective than the multidomain intervention (MeMo-Health-Cog) with placebo in improving insulin resistance by 5%, global cognitive function by 3%, neuropsychological functions, physical performance by 5%, and neuroprotection biomarkers by 5%. Moreover, these effects are expected to be maintained for up to 28 weeks after the intervention is implemented.

Sample size:

The investigators used a sample size calculation for a superiority clinical trial, using the formula of Zong (2009) and Wang (2020), considering alpha less than 0.05, a power of 80%, the investigators considered a superiority of 5% for the intervention group, which was considered clinically significant. the investigators considered differences reported in previous clinically acceptable studies, as well as taking into account the standard deviation. For general cognitive function (MOCA) = 0.20 (0.05), for subjective cognitive function 6 (0.05), Trail Making test part A 0.20 (0.05), Trail Making test part A 0.20 (0.05), verbal learning test (RAVLT-immediate) 0.44 (0.05), verbal test (RAVLT-delayed) 0.58 (0.05), verbal fluency = 0.46 (0.05); GSK-3 beta = 0.40 (0.05), HOMA IR 0.1 (0.05); 4 4 hydroxynonenal 0.12 (0.05), MDA (malondialdehyde) 0.18 (0.05), TNF alpha 2.8 (0.05), TNF alpha effect on RALVT 3.3 (0.05), IL-6 (0.05), IL-1 0.001 (0.3). Taking these parameters into account, the total sample size is 64 participants, but if the investigators add that we need to do a multivariate analysis with at least 3 variables (inflammation, insulin resistance, and oxidative stress) to explain the improvement in patients, the investigators consider that require 50 patients per group, that is, 100 patients in total.

Intervention implementation. The study will be coordinated by the principal investigator of the Epidemiology and Health Services Research Unit of the IMSS in Mexico City, National Medical Center Siglo XXI. The interviews will be conducted in a place assigned by the UMF 4; and the training site. The Education and Research Coordinator at the UMF headquarters will be available to resolve emergencies or any event requiring clinical attention. The experimental group consisted of 60-min sessions conducted three days a week for 24 weeks. Each session will be guided by a health professional with experience in nursing who was previously trained to train with the MeMo-Salud-Cog-4 program. The trainer will apply aerobic exercises and then show different step patterns and ask the participants to observe, memorize and repeat these patterns on the checkered mat. The maximum number of participants per group will be 12.

Motivational strategies. A follow-up system will be an important strategy to prevent dropouts and low adherence to the program. This system will be complemented with motivational phone calls to participants who missed group sessions or who do not take the supplement, as well as to people who missed it due to medical appointments or personal commitments. At the end of the program, the program is extended to complete the sessions at 80%. In addition, the study includes a motivational educational program that consists of group sessions of 10 to 15 minutes to explore topics related to active aging, sports for the elderly, health issues, nutrition and socialization through the exchange of experiences about past events. This program is given before or after the session, depending on the group's decision. The talks have educational material in which the topics are briefly explained on a WEB page and in a book where more information is provided. The instructor, who is a trained health professional, gave the talk through the WEB page and the participant received a book for more information on the topic.

Evaluation. The research will include 3 evaluations: at baseline, 24 weeks, and at 52 weeks. The outcome variables of the study will be measured at each evaluation, as will the covariates. The investigators will measure the participants' adherence to the program, defined as 80%. Finally, the reasons for abandoning the program and poor adherence will be documented. The evaluation will be performed by health professionals with internal medicine and gerontology specialties.

The study included the following covariates: age, biological sex, formal education level, current employment and status (active, retired, volunteer, self-employed), marital status (married, divorced, single, in a common-law relationship, other), current living status (living alone, with wife or husband, living with or without children), comorbidities (hypertension, orthopedic, cardiac, vascular, hepatic or renal disorders), baseline physical activity prior to the study, ideally defined as more than 150 minutes per week of moderate physical activity or more than 75 minutes per week of intense vigorous activity, or an equivalent combination); moderate/intense (less than 149 minutes per week of mild or moderate activity less than 74 minutes of vigorous or intense activity, or its equivalent); and poor (no physical activity, neither moderate nor intense), the presence of the APOE ε4 allele was measured.

Statistical analysis. The researcher will first perform a descriptive analysis of older adults, their results in each assessment, and the distribution of quantitative variables using Kolmogorov-Smirnov as a test to assess normality. Normally distributed variables will be analyzed using means and standard deviations, measurements with free distribution will be presented using median and 25th and 75th percentiles, and categorical variables will be described using frequency and percentage. Second, for each evaluation, the researcher will be able to compare the variables of the groups before and after, the magnitude of the change in these, and their comparisons between groups. For comparisons between groups, the investigators will use the Student t-test (for those with a normal distribution) and the Mann-Whitney U test (for those with a non-normal distribution). The effect of the intervention on the outcome variables will be estimated by measuring the difference in change from baseline to measurements at 24 and 52 weeks, and a comparative analysis of the magnitude of the differences between groups will be performed

The analysis of the difference in means by intervention and control group for continuous and normally distributed response variables will be reported as the mean and standard deviation for variables with normal distribution, and the comparison of the means between t0-t24 weeks and t24 weeks - t52 weeks will be done using the paired t-Student test. For variables without normal distribution, the comparison of medians at t0-t24 weeks and t24 weeks-t52 weeks will be obtained from paired samples using the Wilcoxon test. In both cases, a significant difference will be considered with a value of p less than 0.05. For discrete variables, the difference in proportions will be obtained using the chi-square test, using time zero as reference. The comparison of the effect of the intervention and the control from t0 to t24 weeks for the continuous outcome variables will be estimated by estimating the effects and 95% confidence intervals of the differences in the means ("d") over time using the univariate general linear model, regression analysis, and two-factor analysis of variance (ANOVA). This analysis will include covariates and interactions, contrasting both balanced and unbalanced models, and generating effect estimates with 95% confidence intervals. To check assumptions, a robust analysis of variance will be performed for deviations from normality, ensuring that the assumption of symmetry and homogeneity of variances is met (p more than 0.05). In a second model, a comparison analysis of the effect of the intervention and the control from t24 weeks - t52 weeks will be performed. For variables that do not comply with normality, Generalized Estimating Equations (GEE) will be used, a method suitable for repeated measurements that allows the inclusion of covariates and interactions. The interpretation of the results in favor will be considered when the p value less than 0.05.

For discrete variables, the effect estimation will be performed using logistic regression analysis to estimate the Relative Risk and 95% confidence intervals, reporting raw values and those adjusted for covariates selected based on their clinical or statistical relevance. Models will be obtained for the comparison of the intervention and control t0-t24 weeks and t24-t52 weeks. The interpretation of the results in favor will be considered when the p value less than 0.05.

In both analyses, the interaction of participants with low adherence will be included considering the 25% percentile.

The handling of lost values through multiple imputation or models that handle incomplete data will be considered, ensuring the integrity and validity of longitudinal statistical analyses. The analyses will be performed using Stata V.14.0 software (Stata Corp) and IBM SPSS version 23.

Conditions:

Cognitive Decline Insulin resistance.

Keywords:

cognitive decline multidomain intervention turmeric plus papering.

Study Design

Study Type: Interventional Primary Purpose: Prevention Study Phase: N/A Interventional Study Model: Parallel Assignment A double-blind randomized clinical trial entitled "Mind and Movement: Towards the Cognitive Health of Older Adults 4" will be conducted. The study will include a intervention group and one control group: (1) a multidomain intervention with double-task exercise program with a squared mat led by a coach (a health professional) for 24 weeks plus a turmeric capsule plus black pepper every 12 hours; and a control group included a multidomain intervention with double-task exercise program with a squared mat led by a coach (a health professional) for 24 weeks plus a placebo capsule every 12 hours.

Number of Arms: 2

Masking: Double (Participant, Investigator) To ensure that the groups are balanced regarding varying levels of education, study participants were not stratified and randomly allocated in blocks of four to one of the intervention groups or the control group. An independent researcher who will not participate in the study will use the Random Allocation Software to generate the allocation sequence. Each stratum will have its own seed. This researcher will generate uniform random integers to create the allocation order within each block. She will hold the randomization file on her computer and will give out the allocations of individual participants one at a time to the three groups. The allocations will be concealed from participants and the study staff involved in enrollment and baseline evaluation.

The recruitment and application of the intervention for groups in Care Unit 4 for IMSS.

Allocation: Randomized

Enrollment: 100

Arms and Interventions

Arms

Active Comparator: control group included a multidomain intervention with double-task exercise program with a squared mat led by a coach (a health professional) for 24 weeks plus a placebo capsule every 12 hours.

Assigned Interventions

Mind and Movement for Cognitive Health in the OlderAdult 4" The intervention group will consist of 60-minute training sessions delivered three days a week during a 24-week period. Each session will be guided by a health professional certified to coach SSE. The make-up of each session is: 1) 5 minutes of warm-up; 2) 30 minutes of moderate-to-strong intensity aerobic exercise, 3) 5 minutes of aerobic cool-down, 4) 20 minutes of double -task exercise (mat); and 5) 5 minutes of cool-down stretching (this times does not count as activity) plus a capsule with 500mg of turmeric and 5mg of black Pepper.

Other Names:

Aerobic and stength exercise programa. Double-task exercise by a health professional older adults and their caregivers will participate in the same SSE program led by coach for 24 weeks.

Outcome Measures

Primary Outcome Measure:

1. General Cognitive funtion General cognitive function assessed by the Montreal Cognitive Assessment (MoCA) test on a scale of 0-30 points.

Scores are interpreted as follows: >26 indicates no dementia, 18-26 mild cognitive impairment, 6-10 moderate dementia, and <6 severe dementia. [Time Frame: 0, 24 and 52 weeks]

[Time Frame: 52 weeks] Specific domains of cognitive function Measured through composite scores: Executive function/mental flexibility will be measured with the Trail Making Tests, Part A and Part B. The results for both TMT-A and TMT-B are reported as the number of seconds required to complete a task. Processing speed (using the Digit Symbol Substitution Test) will be measured as the total correct number-symbol matches achieved in 90 seconds. Verbal learning and memory will be assessed through Rey's Auditory Verbal Learning Test (RAVLT) that consists of documenting the number of words remembered from a list of 15 words presented in two separate moments; this test allows evaluation of the RAVLT-Immediate and RAVLT-Percent Forgetting. Verbal fluency (semantic, animal naming, and phonemic) will be measured by using the Controlled Oral Word Association Test and assessed through the total number of words identified by category and letter.

[Time Frame: 0, 24 and 52 weeks]

Metabolic biomarkers, inflammation and oxidative stress damage biomarkers: HOMA-IR, glycosylated hemoglobin, markers of oxidative stress (malondialdehyde, 4-hydroxi-2-nonenal, Thiol groups, carbonyl groups, glutathion peroxidase activity), GSK-3beta, IL-1, IL-6, TNF-alpha.

[Time Frame: 0,12, 24 and 52 weeks]

Cognitive reserve episode. Capacity that enables an individual to cope with and/or recover from the impact of a neural injury or a psychotic [Time Frame: 0 and 52 weeks]

Secondary Outcome Measure:

Usual walking and dual-task gait Usual walking and dual-task gait will be evaluated through motion capture during the six-minute walk test (6MWT), which requires participants to walk back and forth across a 30-metre area at a comfortable pace for six minutes. The fixed distance utilized by 6MWT allows determination of gait speed (i.e., v=d/t); however, this test will also be coupled with infrared stride analysis, which will allow for a more precise evaluation of gait speed, stride length, and stride variability under usual and dual-task conditions. These procedures will provide a number of valid and reliable gait outcomes through the synchronization of mobility data via eight infrared cameras, six force plates, and electromyography.

[Time Frame: 52 weeks]

Quality of life as measured by SF-12 Older adults' health-related quality of life (QoL) will be measured by the short form (SF-12) of the Medical Outcomes Survey questionnaire, comprised of 12 items. Physical and mental scores will be calculated using an algorithm to convert each item response into standardized values according to specific predetermined weights. Summary scores for each component range from 0-100 and are interpreted as low QoL (close to 0) and high QoL (approaching 100).

Cardiovascular biomarkers and endothelial function: MCP-1, ICAM VCAM and Selectin This is the ability of circulating vascular cell adhesion molecule-1 (VCAM-1), endothelial-leukocyte adhesion molecule-1 (E-selectin), and intercellular adhesion molecule-1 (ICAM-1) to serve as molecular markers of atherosclerosis and predictors of incident cardiovascular disease.

[Time Frame: 52 weeks]

ELIGIBILITY:
Inclusion Criteria:

* Minimum Age: 55 Years Maximum Age: 70 Years Sex: All Gender Based: No Accepts Healthy Volunteers: No Criteria: Inclusion criteria.
* 1. With 55-70 years of age.
* 2. They have self-reported cognitive concerns (ie, have answered "yes" to the question: "Do you feel like your memory or thinking skills have gotten worse recently?").
* 3. The participant has insulin resistance measured with HOMA IR index > 2.5.
* 4. They demonstrate functional independence in activities of daily living and instrumental activities of daily living.
* 5. They have symptoms or signs of underlying cognitive dysfunction without a diagnosis of dementia (ie, confirmed by a review of their health records and a Mini Mental State Exam [MMSE] score> 24).
* 6. If the participant are a woman, one year after having gone through menopause.

Exclusion Criteria:

* 1. With depression (score> 15 according to the Center for Epidemiological Studies Depression Scale - Revised [CESD-R]).
* 2. With clinically significant neurological or psychiatric disorders (eg, Parkinson's, schizophrenia).
* 3. With a recent severe cardiovascular event (eg, myocardial infarction, stroke).
* 4. With a major orthopedic condition (eg, severe osteoarthritis).
* 5. With blood pressure that is unsafe for exercise (ie,> 180/100 mmHg or <100/60 mmHg).
* 6. With a severe visual or auditory impairment.
* 7. With an unwillingness to adhere to the intervention schedules.
* 8. Patients with active cancer, who are undergoing chemotherapy, radiotherapy, or other treatments aimed at eradicating cancer and who have been undergoing treatment during the last year.
* 9. Elimination: participants with incomplete data and who have not complied with the intervention by 80%.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Improving insulin resistance by 5%. | 12, 24 y 52 weeks
  The investigadors will measure various parameters of insulin resistance such as glycated hemoglobin, insulin resistance index, and we will measure the improvement of these parameters.
General Cognitive funtion | Time Frame: 0, 24 and 52 weeks
  General cognitive function assessed by the Montreal Cognitive Assessment (MoCA) test on a scale of 0-30 points.
  Scores are interpreted as follows: >26 indicates no dementia, 18-26 mild cognitive impairment, 6-10 moderate dementia.
Specific domains of cognitive function | 0, 24, 52 weeks
  Measured through composite scores: Executive function/mental flexibility will be measured with the Trail Making Tests, Part A and Part B. The results for both TMT-A and TMT-B are reported as the number of seconds required to complete a task. Processing speed (using the Digit Symbol Substitution Test) will be measured as the total correct number-symbol matches achieved in 90 seconds. Verbal learning and memory will be assessed through Rey's Auditory Verbal Learning Test (RAVLT), that consists of documenting the number of words remembered from a list of 15 words presented in two separate moments; this test allows evaluation of the RAVLT-Immediate and RAVLT-Percent Forgetting. Verbal fluency (semantic, animal naming, and phonemic) will be measured by using the Controlled Oral Word Association Test and assessed through the total number of words identified by category and letter.
Oxidative stress. | 0, 12. 24. 52 weeks.
  The investigators will measure several parameters of oxidative stress, including 4-hydroxynonenal (4OH-N), malonaldehyde (MDA), quinones, and glutathione system activity.

SECONDARY OUTCOMES:
Usual walking and dual-task gait | 0 and 52 weeks
  Usual walking and dual-task gait will be evaluated through motion capture during the six-minute walk test (6MWT), which requires participants to walk back and forth across a 30-metre area at a comfortable pace for six minutes. The fixed distance utilized by 6MWT allows determination of gait speed (i.e., v=d/t); however, this test will also be coupled with infrared stride analysis, which will allow for a more precise evaluation of gait speed, stride length, and stride variability under usual and dual-task conditions. These procedures will provide a number of valid and reliable gait outcomes through the synchronization of mobility data via eight infrared cameras, six force plates, and electromyography.
Quality of life as measured by SF-12 | 0 and 52 weeks
  Older adults' health-related quality of life (QoL) will be measured by the short form (SF-12) of the Medical Outcomes Survey questionnaire, comprised of 12 items. Physical and mental scores will be calculated using an algorithm to convert each item response into standardized values according to specific predetermined weights. Summary scores for each component range from 0-100 and are interpreted as low QoL (close to 0) and high QoL (approaching 100).
Cardiovascular biomarkers and endothelial function: MCP-1, ICAM VCAM and Selectin | 0 and 52weeks
  This is the ability of circulating vascular cell adhesion molecule-1 (VCAM-1), endothelial-leukocyte adhesion molecule-1 (E-selectin), and intercellular adhesion molecule-1 (ICAM-1) to serve as molecular markers of atherosclerosis and predictors of incident cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Dubrovna, PhD, Study Director — Instituto Mexicano del Seguro Social
Locations (1):
- Centro Medico Nacional Siglo XXI, unidad de investigación en epidemiología y servicio de salud., Mexico City, Cuauhtémoc, Mexico

IPD SHARING:
Plan to Share IPD: No
Data will be shared on written request

REFERENCES:
- [Background] Hixson JE, Vernier DT. Restriction isotyping of human apolipoprotein E by gene amplification and cleavage with HhaI. J Lipid Res. 1990 Mar;31(3):545-8. PMID 2341813
- [Background] Raulin AC, Doss SV, Trottier ZA, Ikezu TC, Bu G, Liu CC. ApoE in Alzheimer's disease: pathophysiology and therapeutic strategies. Mol Neurodegener. 2022 Nov 8;17(1):72. doi: 10.1186/s13024-022-00574-4. PMID 36348357
- [Background] Custodia A, Aramburu-Nunez M, Rodriguez-Arrizabalaga M, Pias-Peleteiro JM, Vazquez-Vazquez L, Camino-Castineiras J, Aldrey JM, Castillo J, Ouro A, Sobrino T, Romaus-Sanjurjo D. Biomarkers Assessing Endothelial Dysfunction in Alzheimer's Disease. Cells. 2023 Mar 22;12(6):962. doi: 10.3390/cells12060962. PMID 36980302
- [Background] Johnson FK, Peyton KJ, Liu XM, Azam MA, Shebib AR, Johnson RA, Durante W. Arginase promotes endothelial dysfunction and hypertension in obese rats. Obesity (Silver Spring). 2015 Feb;23(2):383-90. doi: 10.1002/oby.20969. Epub 2014 Dec 31. PMID 25557182
- [Background] Gieseg SP, Simpson JA, Charlton TS, Duncan MW, Dean RT. Protein-bound 3,4-dihydroxyphenylalanine is a major reductant formed during hydroxyl radical damage to proteins. Biochemistry. 1993 May 11;32(18):4780-6. doi: 10.1021/bi00069a012. PMID 8387814
- [Background] Dean RT, Gieseg S, Davies MJ. Reactive species and their accumulation on radical-damaged proteins. Trends Biochem Sci. 1993 Nov;18(11):437-41. doi: 10.1016/0968-0004(93)90145-d. PMID 8291091
- [Background] Garcia-Blanco A, Baquero M, Vento M, Gil E, Bataller L, Chafer-Pericas C. Potential oxidative stress biomarkers of mild cognitive impairment due to Alzheimer disease. J Neurol Sci. 2017 Feb 15;373:295-302. doi: 10.1016/j.jns.2017.01.020. Epub 2017 Jan 7. PMID 28131209
- [Background] Mandal PK, Saharan S, Khan SA, James M. Apps for Dementia Screening: A Cost-effective and Portable Solution. J Alzheimers Dis. 2015;47(4):869-72. doi: 10.3233/JAD-150255. No abstract available. PMID 26401765
- [Background] Malek-Ahmadi M, Small BJ, Raj A. The diagnostic value of controlled oral word association test-FAS and category fluency in single-domain amnestic mild cognitive impairment. Dement Geriatr Cogn Disord. 2011;32(4):235-40. doi: 10.1159/000334525. Epub 2011 Dec 8. PMID 22156335
- [Background] Moradi E, Hallikainen I, Hanninen T, Tohka J; Alzheimer's Disease Neuroimaging Initiative. Rey's Auditory Verbal Learning Test scores can be predicted from whole brain MRI in Alzheimer's disease. Neuroimage Clin. 2016 Dec 18;13:415-427. doi: 10.1016/j.nicl.2016.12.011. eCollection 2017. PMID 28116234
- [Background] Rosano C, Perera S, Inzitari M, Newman AB, Longstreth WT, Studenski S. Digit Symbol Substitution test and future clinical and subclinical disorders of cognition, mobility and mood in older adults. Age Ageing. 2016 Sep;45(5):688-95. doi: 10.1093/ageing/afw116. Epub 2016 Jul 4. PMID 27496932
- [Background] Gaudino EA, Geisler MW, Squires NK. Construct validity in the Trail Making Test: what makes Part B harder? J Clin Exp Neuropsychol. 1995 Aug;17(4):529-35. doi: 10.1080/01688639508405143. PMID 7593473
- [Background] Aguilar-Navarro SG, Mimenza-Alvarado AJ, Palacios-Garcia AA, Samudio-Cruz A, Gutierrez-Gutierrez LA, Avila-Funes JA. Validity and Reliability of the Spanish Version of the Montreal Cognitive Assessment (MoCA) for the Detection of Cognitive Impairment in Mexico. Rev Colomb Psiquiatr (Engl Ed). 2018 Oct-Dec;47(4):237-243. doi: 10.1016/j.rcp.2017.05.003. Epub 2017 Jul 29. English, Spanish. PMID 30286846
- [Background] Saghaei M. Random allocation software for parallel group randomized trials. BMC Med Res Methodol. 2004 Nov 9;4:26. doi: 10.1186/1471-2288-4-26. PMID 15535880
- [Background] Kohout FJ, Berkman LF, Evans DA, Cornoni-Huntley J. Two shorter forms of the CES-D (Center for Epidemiological Studies Depression) depression symptoms index. J Aging Health. 1993 May;5(2):179-93. doi: 10.1177/089826439300500202. PMID 10125443
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Kelly ME, Loughrey D, Lawlor BA, Robertson IH, Walsh C, Brennan S. The impact of cognitive training and mental stimulation on cognitive and everyday functioning of healthy older adults: a systematic review and meta-analysis. Ageing Res Rev. 2014 May;15:28-43. doi: 10.1016/j.arr.2014.02.004. Epub 2014 Mar 4. PMID 24607830
- [Background] Willis SL, Tennstedt SL, Marsiske M, Ball K, Elias J, Koepke KM, Morris JN, Rebok GW, Unverzagt FW, Stoddard AM, Wright E; ACTIVE Study Group. Long-term effects of cognitive training on everyday functional outcomes in older adults. JAMA. 2006 Dec 20;296(23):2805-14. doi: 10.1001/jama.296.23.2805. PMID 17179457
- [Background] Licastro F, Pedrini S, Caputo L, Annoni G, Davis LJ, Ferri C, Casadei V, Grimaldi LM. Increased plasma levels of interleukin-1, interleukin-6 and alpha-1-antichymotrypsin in patients with Alzheimer's disease: peripheral inflammation or signals from the brain? J Neuroimmunol. 2000 Feb 1;103(1):97-102. doi: 10.1016/s0165-5728(99)00226-x. PMID 10674995
- [Background] Lyra E Silva NM, Goncalves RA, Pascoal TA, Lima-Filho RAS, Resende EPF, Vieira ELM, Teixeira AL, de Souza LC, Peny JA, Fortuna JTS, Furigo IC, Hashiguchi D, Miya-Coreixas VS, Clarke JR, Abisambra JF, Longo BM, Donato J Jr, Fraser PE, Rosa-Neto P, Caramelli P, Ferreira ST, De Felice FG. Pro-inflammatory interleukin-6 signaling links cognitive impairments and peripheral metabolic alterations in Alzheimer's disease. Transl Psychiatry. 2021 Apr 28;11(1):251. doi: 10.1038/s41398-021-01349-z. PMID 33911072
- [Background] Windham BG, Simpson BN, Lirette S, Bridges J, Bielak L, Peyser PA, Kullo I, Turner S, Griswold ME, Mosley TH. Associations between inflammation and cognitive function in African Americans and European Americans. J Am Geriatr Soc. 2014 Dec;62(12):2303-10. doi: 10.1111/jgs.13165. PMID 25516026
- [Background] Xing YW, Liu KZ. Azithromycin inhibited oxidative stress and apoptosis of high glucose-induced podocytes by inhibiting STAT1 pathway. Drug Dev Res. 2021 Nov;82(7):990-998. doi: 10.1002/ddr.21801. Epub 2021 Mar 2. PMID 33655586
- [Background] Markesbery WR. Oxidative stress hypothesis in Alzheimer's disease. Free Radic Biol Med. 1997;23(1):134-47. doi: 10.1016/s0891-5849(96)00629-6. PMID 9165306
- [Background] Gill DP, Gregory MA, Zou G, Liu-Ambrose T, Shigematsu R, Hachinski V, Fitzgerald C, Petrella RJ. The Healthy Mind, Healthy Mobility Trial: A Novel Exercise Program for Older Adults. Med Sci Sports Exerc. 2016 Feb;48(2):297-306. doi: 10.1249/MSS.0000000000000758. PMID 26285025
- [Background] Abner EL, Kryscio RJ, Caban-Holt AM, Schmitt FA. Baseline subjective memory complaints associate with increased risk of incident dementia: the PREADVISE trial. J Prev Alzheimers Dis. 2015 Mar;2(1):11-16. doi: 10.14283/jpad.2015.37. PMID 26180776
- [Background] Wang X, Ji X. Sample Size Estimation in Clinical Research: From Randomized Controlled Trials to Observational Studies. Chest. 2020 Jul;158(1S):S12-S20. doi: 10.1016/j.chest.2020.03.010. PMID 32658647
- [Background] Zhong B. How to calculate sample size in randomized controlled trial? J Thorac Dis. 2009 Dec;1(1):51-4. PMID 22263004
- [Background] Camacho-Ruiz J, V A, Rendon-Macias ME, Bernabe-Garcia M, Gonzalez-Bautista E, Manuel-Apolinar L, Basurto-Acevedo L, Orihuela-Rodriguez O, M Ruiz-Batalla J, Rojas-Rubio B, Olivares-Santos RA, Paredes-Manjarrez C, Sanchez-Arenas R. [Cognitive function groups in older people and risk factors]. Rev Med Inst Mex Seguro Soc. 2024 May 6;62(3):1-11. doi: 10.5281/zenodo.10998801. Spanish. PMID 39528344
- [Background] Mimenza-Alvarado A, Aguilar-Navarro SG, Yeverino-Castro S, Mendoza-Franco C, Avila-Funes JA, Roman GC. Neuroimaging Characteristics of Small-Vessel Disease in Older Adults with Normal Cognition, Mild Cognitive Impairment, and Alzheimer Disease. Dement Geriatr Cogn Dis Extra. 2018 May 16;8(2):199-206. doi: 10.1159/000488705. eCollection 2018 May-Aug. PMID 29928288
- [Background] Zahedipour F, Hosseini SA, Sathyapalan T, Majeed M, Jamialahmadi T, Al-Rasadi K, Banach M, Sahebkar A. Potential effects of curcumin in the treatment of COVID-19 infection. Phytother Res. 2020 Nov;34(11):2911-2920. doi: 10.1002/ptr.6738. Epub 2020 Jun 23. PMID 32430996
- [Background] Hoppe JB, Haag M, Whalley BJ, Salbego CG, Cimarosti H. Curcumin protects organotypic hippocampal slice cultures from Abeta1-42-induced synaptic toxicity. Toxicol In Vitro. 2013 Dec;27(8):2325-30. doi: 10.1016/j.tiv.2013.10.002. Epub 2013 Oct 14. PMID 24134851
- [Background] Khandia R, Viswanathan N, Singhal S, Alqahtani T, Almikhlafi MA, Simonov AN, Ashraf GM. Ameliorative Effects of Phytomedicines on Alzheimer's Patients. Curr Alzheimer Res. 2022;19(6):420-439. doi: 10.2174/1567205019666220610155608. PMID 35692129
- [Background] Berry A, Collacchi B, Masella R, Vari R, Cirulli F. Curcuma Longa, the "Golden Spice" to Counteract Neuroinflammaging and Cognitive Decline-What Have We Learned and What Needs to Be Done. Nutrients. 2021 Apr 30;13(5):1519. doi: 10.3390/nu13051519. PMID 33946356
- [Background] Randino R, Grimaldi M, Persico M, De Santis A, Cini E, Cabri W, Riva A, D'Errico G, Fattorusso C, D'Ursi AM, Rodriquez M. Investigating the Neuroprotective Effects of Turmeric Extract: Structural Interactions of beta-Amyloid Peptide with Single Curcuminoids. Sci Rep. 2016 Dec 22;6:38846. doi: 10.1038/srep38846. PMID 28004737
- [Background] Chainoglou E, Hadjipavlou-Litina D. Curcumin in Health and Diseases: Alzheimer's Disease and Curcumin Analogues, Derivatives, and Hybrids. Int J Mol Sci. 2020 Mar 13;21(6):1975. doi: 10.3390/ijms21061975. PMID 32183162
- [Background] Kocaadam B, Sanlier N. Curcumin, an active component of turmeric (Curcuma longa), and its effects on health. Crit Rev Food Sci Nutr. 2017 Sep 2;57(13):2889-2895. doi: 10.1080/10408398.2015.1077195. PMID 26528921
- [Background] Thota RN, Rosato JI, Dias CB, Burrows TL, Martins RN, Garg ML. Dietary Supplementation with Curcumin Reduce Circulating Levels of Glycogen Synthase Kinase-3beta and Islet Amyloid Polypeptide in Adults with High Risk of Type 2 Diabetes and Alzheimer's Disease. Nutrients. 2020 Apr 9;12(4):1032. doi: 10.3390/nu12041032. PMID 32283762
- [Background] Hewlings SJ, Kalman DS. Curcumin: A Review of Its Effects on Human Health. Foods. 2017 Oct 22;6(10):92. doi: 10.3390/foods6100092. PMID 29065496
- [Background] Anand P, Kunnumakkara AB, Newman RA, Aggarwal BB. Bioavailability of curcumin: problems and promises. Mol Pharm. 2007 Nov-Dec;4(6):807-18. doi: 10.1021/mp700113r. Epub 2007 Nov 14. PMID 17999464
- [Background] Ryu EK, Choe YS, Lee KH, Choi Y, Kim BT. Curcumin and dehydrozingerone derivatives: synthesis, radiolabeling, and evaluation for beta-amyloid plaque imaging. J Med Chem. 2006 Oct 5;49(20):6111-9. doi: 10.1021/jm0607193. PMID 17004725
- [Background] Murakami M, Ikeda Y, Nakagawa Y, Tsuji A, Kitagishi Y, Matsuda S. Special bioactive compounds and functional foods may exhibit neuroprotective effects in patients with dementia (Review). Biomed Rep. 2020 Aug;13(2):1. doi: 10.3892/br.2020.1310. Epub 2020 Jun 2. PMID 32509304
- [Background] Ferrari CK. Functional foods and physical activities in health promotion of aging people. Maturitas. 2007 Dec 20;58(4):327-39. doi: 10.1016/j.maturitas.2007.09.011. Epub 2007 Nov 5. PMID 17980978
- [Background] Janelidze S, Mattsson N, Stomrud E, Lindberg O, Palmqvist S, Zetterberg H, Blennow K, Hansson O. CSF biomarkers of neuroinflammation and cerebrovascular dysfunction in early Alzheimer disease. Neurology. 2018 Aug 28;91(9):e867-e877. doi: 10.1212/WNL.0000000000006082. Epub 2018 Jul 27. PMID 30054439
- [Background] Qiu S, Cai X, Liu J, Yang B, Zugel M, Steinacker JM, Sun Z, Schumann U. Association between circulating cell adhesion molecules and risk of type 2 diabetes: A meta-analysis. Atherosclerosis. 2019 Aug;287:147-154. doi: 10.1016/j.atherosclerosis.2019.06.908. Epub 2019 Jun 20. PMID 31280040
- [Background] Meigs JB, Hu FB, Rifai N, Manson JE. Biomarkers of endothelial dysfunction and risk of type 2 diabetes mellitus. JAMA. 2004 Apr 28;291(16):1978-86. doi: 10.1001/jama.291.16.1978. PMID 15113816
- [Background] Toledo JB, Arnold SE, Raible K, Brettschneider J, Xie SX, Grossman M, Monsell SE, Kukull WA, Trojanowski JQ. Contribution of cerebrovascular disease in autopsy confirmed neurodegenerative disease cases in the National Alzheimer's Coordinating Centre. Brain. 2013 Sep;136(Pt 9):2697-706. doi: 10.1093/brain/awt188. Epub 2013 Jul 10. PMID 23842566
- [Background] Pedersen BK. Physical activity and muscle-brain crosstalk. Nat Rev Endocrinol. 2019 Jul;15(7):383-392. doi: 10.1038/s41574-019-0174-x. PMID 30837717
- [Background] Tumminia A, Vinciguerra F, Parisi M, Frittitta L. Type 2 Diabetes Mellitus and Alzheimer's Disease: Role of Insulin Signalling and Therapeutic Implications. Int J Mol Sci. 2018 Oct 24;19(11):3306. doi: 10.3390/ijms19113306. PMID 30355995
- [Background] Hoppe JB, Coradini K, Frozza RL, Oliveira CM, Meneghetti AB, Bernardi A, Pires ES, Beck RC, Salbego CG. Free and nanoencapsulated curcumin suppress beta-amyloid-induced cognitive impairments in rats: involvement of BDNF and Akt/GSK-3beta signaling pathway. Neurobiol Learn Mem. 2013 Nov;106:134-44. doi: 10.1016/j.nlm.2013.08.001. Epub 2013 Aug 14. PMID 23954730
- [Background] Liang LL, He MF, Zhou PP, Pan SK, Liu DW, Liu ZS. GSK3beta: A ray of hope for the treatment of diabetic kidney disease. FASEB J. 2024 Feb 15;38(3):e23458. doi: 10.1096/fj.202302160R. PMID 38315453
- [Background] Wang YJ, Ren QG, Gong WG, Wu D, Tang X, Li XL, Wu FF, Bai F, Xu L, Zhang ZJ. Escitalopram attenuates beta-amyloid-induced tau hyperphosphorylation in primary hippocampal neurons through the 5-HT1A receptor mediated Akt/GSK-3beta pathway. Oncotarget. 2016 Mar 22;7(12):13328-39. doi: 10.18632/oncotarget.7798. PMID 26950279
- [Background] Li X, Jope RS. Is glycogen synthase kinase-3 a central modulator in mood regulation? Neuropsychopharmacology. 2010 Oct;35(11):2143-54. doi: 10.1038/npp.2010.105. Epub 2010 Jul 28. PMID 20668436
- [Background] Jia YR, Guo ZQ, Guo Q, Wang XC. Glycogen Synthase Kinase-3beta, NLRP3 Inflammasome, and Alzheimer's Disease. Curr Med Sci. 2023 Oct;43(5):847-854. doi: 10.1007/s11596-023-2788-4. Epub 2023 Sep 18. PMID 37721665
- [Background] Rafii MS, Aisen PS. Detection and treatment of Alzheimer's disease in its preclinical stage. Nat Aging. 2023 May;3(5):520-531. doi: 10.1038/s43587-023-00410-4. Epub 2023 May 18. PMID 37202518
- [Background] Mandal PK, Saharan S, Tripathi M, Murari G. Brain glutathione levels--a novel biomarker for mild cognitive impairment and Alzheimer's disease. Biol Psychiatry. 2015 Nov 15;78(10):702-10. doi: 10.1016/j.biopsych.2015.04.005. Epub 2015 Apr 14. PMID 26003861
- [Background] Bradley-Whitman MA, Lovell MA. Biomarkers of lipid peroxidation in Alzheimer disease (AD): an update. Arch Toxicol. 2015 Jul;89(7):1035-44. doi: 10.1007/s00204-015-1517-6. Epub 2015 Apr 18. PMID 25895140
- [Background] Gigase FAJ, Smith E, Collins B, Moore K, Snijders GJLJ, Katz D, Bergink V, Perez-Rodriquez MM, De Witte LD. The association between inflammatory markers in blood and cerebrospinal fluid: a systematic review and meta-analysis. Mol Psychiatry. 2023 Apr;28(4):1502-1515. doi: 10.1038/s41380-023-01976-6. Epub 2023 Apr 13. PMID 37055513
- [Background] Albar NY, Hassaballa H, Shikh H, Albar Y, Ibrahim AS, Mousa AH, Alshanberi AM, Elgebaly A, Bahbah EI. The interaction between insulin resistance and Alzheimer's disease: a review article. Postgrad Med. 2024 May;136(4):377-395. doi: 10.1080/00325481.2024.2360887. Epub 2024 Jun 4. PMID 38804907
- [Background] Sedzikowska A, Szablewski L. Insulin and Insulin Resistance in Alzheimer's Disease. Int J Mol Sci. 2021 Sep 15;22(18):9987. doi: 10.3390/ijms22189987. PMID 34576151
- [Background] Leng F, Edison P. Neuroinflammation and microglial activation in Alzheimer disease: where do we go from here? Nat Rev Neurol. 2021 Mar;17(3):157-172. doi: 10.1038/s41582-020-00435-y. Epub 2020 Dec 14. PMID 33318676
- [Background] Li H, Ren J, Li Y, Wu Q, Wei J. Oxidative stress: The nexus of obesity and cognitive dysfunction in diabetes. Front Endocrinol (Lausanne). 2023 Apr 3;14:1134025. doi: 10.3389/fendo.2023.1134025. eCollection 2023. PMID 37077347
- [Background] Arellano-Campos O, Gomez-Velasco DV, Bello-Chavolla OY, Cruz-Bautista I, Melgarejo-Hernandez MA, Munoz-Hernandez L, Guillen LE, Garduno-Garcia JJ, Alvirde U, Ono-Yoshikawa Y, Choza-Romero R, Sauque-Reyna L, Garay-Sevilla ME, Malacara-Hernandez JM, Tusie-Luna MT, Gutierrez-Robledo LM, Gomez-Perez FJ, Rojas R, Aguilar-Salinas CA. Development and validation of a predictive model for incident type 2 diabetes in middle-aged Mexican adults: the metabolic syndrome cohort. BMC Endocr Disord. 2019 Apr 28;19(1):41. doi: 10.1186/s12902-019-0361-8. PMID 31030672
- [Background] Rojas R, Aguilar-Salinas CA, Jimenez-Corona A, Shamah-Levy T, Rauda J, Avila-Burgos L, Villalpando S, Ponce EL. Metabolic syndrome in Mexican adults: results from the National Health and Nutrition Survey 2006. Salud Publica Mex. 2010;52 Suppl 1:S11-8. doi: 10.1590/s0036-36342010000700004. PMID 20585723
- [Background] Gastaldelli A. Measuring and estimating insulin resistance in clinical and research settings. Obesity (Silver Spring). 2022 Aug;30(8):1549-1563. doi: 10.1002/oby.23503. PMID 35894085
- [Background] Haeusler RA, McGraw TE, Accili D. Biochemical and cellular properties of insulin receptor signalling. Nat Rev Mol Cell Biol. 2018 Jan;19(1):31-44. doi: 10.1038/nrm.2017.89. Epub 2017 Oct 4. PMID 28974775
- [Background] Rodriguez-Colman MJ, Dansen TB, Burgering BMT. FOXO transcription factors as mediators of stress adaptation. Nat Rev Mol Cell Biol. 2024 Jan;25(1):46-64. doi: 10.1038/s41580-023-00649-0. Epub 2023 Sep 14. PMID 37710009
- [Background] Lennicke C, Cocheme HM. Redox metabolism: ROS as specific molecular regulators of cell signaling and function. Mol Cell. 2021 Sep 16;81(18):3691-3707. doi: 10.1016/j.molcel.2021.08.018. PMID 34547234
- [Background] James DE, Stockli J, Birnbaum MJ. The aetiology and molecular landscape of insulin resistance. Nat Rev Mol Cell Biol. 2021 Nov;22(11):751-771. doi: 10.1038/s41580-021-00390-6. Epub 2021 Jul 20. PMID 34285405
- [Background] Yang Q, Vijayakumar A, Kahn BB. Metabolites as regulators of insulin sensitivity and metabolism. Nat Rev Mol Cell Biol. 2018 Oct;19(10):654-672. doi: 10.1038/s41580-018-0044-8. PMID 30104701
- [Background] DeFronzo RA, Ferrannini E, Groop L, Henry RR, Herman WH, Holst JJ, Hu FB, Kahn CR, Raz I, Shulman GI, Simonson DC, Testa MA, Weiss R. Type 2 diabetes mellitus. Nat Rev Dis Primers. 2015 Jul 23;1:15019. doi: 10.1038/nrdp.2015.19. PMID 27189025
- [Background] Biessels GJ, Despa F. Cognitive decline and dementia in diabetes mellitus: mechanisms and clinical implications. Nat Rev Endocrinol. 2018 Oct;14(10):591-604. doi: 10.1038/s41574-018-0048-7. PMID 30022099
- [Background] Shigematsu R, Okura T, Nakagaichi M, Tanaka K, Sakai T, Kitazumi S, Rantanen T. Square-stepping exercise and fall risk factors in older adults: a single-blind, randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2008 Jan;63(1):76-82. doi: 10.1093/gerona/63.1.76. PMID 18245764
- [Background] Shigematsu R, Okura T. A novel exercise for improving lower-extremity functional fitness in the elderly. Aging Clin Exp Res. 2006 Jun;18(3):242-8. doi: 10.1007/BF03324655. PMID 16804371
- [Background] Sanchez-Arenas R, Doubova SV, Bernabe-Garcia M, Gregory MA, Mejia-Alonso LA, Orihuela-Rodriguez O, Paredes-Manjarrez C, Colin-Martinez T, Mujica-Morales I, Grijalva-Otero I, Basurto-Acevedo L, Manuel-Apolinar L, Cuadros-Moreno J, Bernal-Diaz A, Shigematsu R. Double-task exercise programmes to strengthen cognitive and vascular health in older adults at risk of cognitive decline: protocol for a randomised clinical trial. BMJ Open. 2020 Dec 30;10(12):e039723. doi: 10.1136/bmjopen-2020-039723. PMID 33380479
- [Background] Wahl D, Cavalier AN, LaRocca TJ. Novel Strategies for Healthy Brain Aging. Exerc Sport Sci Rev. 2021 Apr 1;49(2):115-125. doi: 10.1249/JES.0000000000000242. PMID 33739944
- [Background] Stillman CM, Esteban-Cornejo I, Brown B, Bender CM, Erickson KI. Effects of Exercise on Brain and Cognition Across Age Groups and Health States. Trends Neurosci. 2020 Jul;43(7):533-543. doi: 10.1016/j.tins.2020.04.010. Epub 2020 May 11. PMID 32409017
- [Background] Piercy KL, Troiano RP, Ballard RM, Carlson SA, Fulton JE, Galuska DA, George SM, Olson RD. The Physical Activity Guidelines for Americans. JAMA. 2018 Nov 20;320(19):2020-2028. doi: 10.1001/jama.2018.14854. PMID 30418471
- [Background] Ross R, Chaput JP, Giangregorio LM, Janssen I, Saunders TJ, Kho ME, Poitras VJ, Tomasone JR, El-Kotob R, McLaughlin EC, Duggan M, Carrier J, Carson V, Chastin SF, Latimer-Cheung AE, Chulak-Bozzer T, Faulkner G, Flood SM, Gazendam MK, Healy GN, Katzmarzyk PT, Kennedy W, Lane KN, Lorbergs A, Maclaren K, Marr S, Powell KE, Rhodes RE, Ross-White A, Welsh F, Willumsen J, Tremblay MS. Canadian 24-Hour Movement Guidelines for Adults aged 18-64 years and Adults aged 65 years or older: an integration of physical activity, sedentary behaviour, and sleep. Appl Physiol Nutr Metab. 2020 Oct;45(10 (Suppl. 2)):S57-S102. doi: 10.1139/apnm-2020-0467. PMID 33054332
- [Background] Boa Sorte Silva NC, Gregory MA, Gill DP, Petrella RJ. Multiple-modality exercise and mind-motor training to improve cardiovascular health and fitness in older adults at risk for cognitive impairment: A randomized controlled trial. Arch Gerontol Geriatr. 2017 Jan-Feb;68:149-160. doi: 10.1016/j.archger.2016.10.009. Epub 2016 Oct 24. PMID 27810663
- [Background] Boa Sorte Silva NC, Gill DP, Gregory MA, Bocti J, Petrella RJ. Multiple-modality exercise and mind-motor training to improve mobility in older adults: A randomized controlled trial. Exp Gerontol. 2018 Mar;103:17-26. doi: 10.1016/j.exger.2017.12.011. Epub 2017 Dec 17. PMID 29262308
- [Background] Andrieu S, Coley N, Lovestone S, Aisen PS, Vellas B. Prevention of sporadic Alzheimer's disease: lessons learned from clinical trials and future directions. Lancet Neurol. 2015 Sep;14(9):926-944. doi: 10.1016/S1474-4422(15)00153-2. Epub 2015 Jul 23. PMID 26213339
- [Background] Jessen F, Amariglio RE, Buckley RF, van der Flier WM, Han Y, Molinuevo JL, Rabin L, Rentz DM, Rodriguez-Gomez O, Saykin AJ, Sikkes SAM, Smart CM, Wolfsgruber S, Wagner M. The characterisation of subjective cognitive decline. Lancet Neurol. 2020 Mar;19(3):271-278. doi: 10.1016/S1474-4422(19)30368-0. Epub 2020 Jan 17. PMID 31958406
- [Background] Dubois B, Hampel H, Feldman HH, Scheltens P, Aisen P, Andrieu S, Bakardjian H, Benali H, Bertram L, Blennow K, Broich K, Cavedo E, Crutch S, Dartigues JF, Duyckaerts C, Epelbaum S, Frisoni GB, Gauthier S, Genthon R, Gouw AA, Habert MO, Holtzman DM, Kivipelto M, Lista S, Molinuevo JL, O'Bryant SE, Rabinovici GD, Rowe C, Salloway S, Schneider LS, Sperling R, Teichmann M, Carrillo MC, Cummings J, Jack CR Jr; Proceedings of the Meeting of the International Working Group (IWG) and the American Alzheimer's Association on "The Preclinical State of AD"; July 23, 2015; Washington DC, USA. Preclinical Alzheimer's disease: Definition, natural history, and diagnostic criteria. Alzheimers Dement. 2016 Mar;12(3):292-323. doi: 10.1016/j.jalz.2016.02.002. PMID 27012484
- [Background] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Background] Frisoni GB, Altomare D, Ribaldi F, Villain N, Brayne C, Mukadam N, Abramowicz M, Barkhof F, Berthier M, Bieler-Aeschlimann M, Blennow K, Brioschi Guevara A, Carrera E, Chetelat G, Csajka C, Demonet JF, Dodich A, Garibotto V, Georges J, Hurst S, Jessen F, Kivipelto M, Llewellyn DJ, McWhirter L, Milne R, Minguillon C, Miniussi C, Molinuevo JL, Nilsson PM, Noyce A, Ranson JM, Grau-Rivera O, Schott JM, Solomon A, Stephen R, van der Flier W, van Duijn C, Vellas B, Visser LNC, Cummings JL, Scheltens P, Ritchie C, Dubois B. Dementia prevention in memory clinics: recommendations from the European task force for brain health services. Lancet Reg Health Eur. 2023 Jan 31;26:100576. doi: 10.1016/j.lanepe.2022.100576. eCollection 2023 Mar. PMID 36895446
- [Background] Ribeiro F, Teixeira-Santos AC, Caramelli P, Leist AK. Prevalence of dementia in Latin America and Caribbean countries: Systematic review and meta-analyses exploring age, sex, rurality, and education as possible determinants. Ageing Res Rev. 2022 Nov;81:101703. doi: 10.1016/j.arr.2022.101703. Epub 2022 Aug 3. PMID 35931410
- [Background] Mukadam N, Sommerlad A, Huntley J, Livingston G. Population attributable fractions for risk factors for dementia in low-income and middle-income countries: an analysis using cross-sectional survey data. Lancet Glob Health. 2019 May;7(5):e596-e603. doi: 10.1016/S2214-109X(19)30074-9. PMID 31000129
- [Background] Ganguli M, Albanese E, Seshadri S, Bennett DA, Lyketsos C, Kukull WA, Skoog I, Hendrie HC. Population Neuroscience: Dementia Epidemiology Serving Precision Medicine and Population Health. Alzheimer Dis Assoc Disord. 2018 Jan-Mar;32(1):1-9. doi: 10.1097/WAD.0000000000000237. PMID 29319603
- [Background] Altomare D, Molinuevo JL, Ritchie C, Ribaldi F, Carrera E, Dubois B, Jessen F, McWhirter L, Scheltens P, van der Flier WM, Vellas B, Demonet JF, Frisoni GB; European Task Force for Brain Health Services. Brain Health Services: organization, structure, and challenges for implementation. A user manual for Brain Health Services-part 1 of 6. Alzheimers Res Ther. 2021 Oct 11;13(1):168. doi: 10.1186/s13195-021-00827-2. PMID 34635163